CLINICAL TRIAL: NCT04920149
Title: Mesalamine for Colorectal Cancer Prevention Program in Lynch Syndrome
Acronym: MesaCAPP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ann-Sofie Backman (Other)
Collaborators: The Swedish Research Council (Other Government); Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Ann-Sofie Backman, Consultant gastroenterology, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MesaCAPP
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Lynch Syndrome; Colon Cancer; Colon Neoplasm
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Colonic Neoplasms | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesalamine (Experimental): Mesalamine (Mesalazine, Pentasa sachet, 5-ASA) 2 g once daily for 2 years.
  Interventions: Drug: Mesalamine
- Placebo (Placebo Comparator): Placebo for Mesalamine (Mesalazine, Pentasa sachet, 5-ASA) 2 g once daily for 2 years.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mesalamine — The IMP will be supplied as sachets with slow-releasing granules.
  Other Names: Mesalazine; Pentasa sachet; 5-ASA
  Arms: Mesalamine
Drug: Placebo — The IMP will be supplied as sachets with slow-releasing granules.
  Arms: Placebo

SUMMARY:
Multicenter, multinational, randomized, 2-arm, double-blind, phase II clinical study with 2000mg mesalamine, or placebo for prevention of colorectal neoplasia in Lynch Syndrome patients during and following daily intake for 2 years.

DETAILED DESCRIPTION:
This is a multicenter, multinational, randomized, 2-arm, double-blind, phase II clinical study with 2000mg mesalamine (5-ASA) or placebo in LS patients for a 2-year treatment. 260 tumor free carriers of a known genetic mutation in a major MMR gene (including patients in which the polyps are endoscopically removed) will be randomized 1:1 to receive 2000mg mesalamine or placebo. Patients will be identified through local or national registries and through collaboration with sites. Tumor free patients, assessed by white light high resolution colonoscopy, will be randomized to the study. Blood and stool samples will be collected for analysis of microbiota, ctDNA and potential biomarkers. Biopsies of the normal tissue of ascending colon and rectum will be taken at the first and the last colonoscopy.

The aim of the study is to investigate the effect of regular treatment with mesalamine (5-ASA) on the occurrence of any colorectal neoplasia, tumor multiplicity (the number of detected adenomas/carcinomas) and tumor progression in LS patients.

Tumor multiplicity and tumor progression (severity of the neoplastic lesions) will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Proven tumor-free (including patients in which the polyps are removed endoscopically) carriers of a germline pathologic mutation in one of the MMR genes including MLH1, MSH2 (including EpCAM) and MSH6
* Male or female subjects with the age of 30 years or older
* Females who have been post-menopausal more than one (1) year or females of childbearing potential using a highly efficient method of contraception with less than 1% failure rate (i.e. oral hormonal contraceptives, hormone implants, hormone injections, sterilization, hormonal or copper intrauterine device, sterilized/vasectomized partner, or diaphragm in combination with a condom, spermicide or birth control pills) or should agree to abstain from heterosexual activity during treatment period. Females of childbearing potential must have a negative pregnancy test at screening and before randomization.
* Signed written informed consent prior to inclusion in the study

Exclusion Criteria:

* Presence of colorectal endoscopically non-removable benign neoplasia (patient can be included if the adenoma is removed)
* Carriers of germline mutations in PMS2
* Patients with history of stage 3 and 4 CRC are excluded
* Presence of metastatic disease
* Regular use of aspirin/ASA: daily use of ≥100mg in more than 3 continuous months within the last year
* Regular use of NSAIDs or COX-2 inhibitors: daily use in more than 3 continuous months within the last year
* Hypersensitivity to 5-ASA
* Patients after any subtotal or total colectomy
* Colorectal surgery within the previous 6 months
* Unwillingness to participate or who is considered incompetent to give an informed consent
* Pregnant or breastfeeding women
* Participation in another clinical study investigating another IMP within 1 month prior to screening
* Renal insufficiency (GFR <30ml/min/1.73m2)
* Severe liver disease or liver failure (elevation of liver enzymes above 3xULN)
* Current or history of serious psychiatric disorder or alcohol/drug abuse that in the opinion of the investigator may impact the assessment of IMP safety and efficacy or protocol adherence
* Prior history of myocarditis or pericarditis. Other severe acute or chronic medical condition such as severe chronic lung (COPD, including asthma, kidney and heart diseases) or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or ability to comply with study procedures, investigational product administration and, in the judgment of the investigator, would make the subject inappropriate for entry into this study

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2032-09-30 (Estimated); Study Completion 2045-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in the occurrence of any colorectal neoplasia in LS patients | End of treatment at 24 months +/- 1 month
  Occurrence of any colorectal neoplasia (both benign and malignant tumors) between groups is described by absolute frequencies and percentages.
Change in the occurrence of any colorectal neoplasia in LS patients | End of study at year 6 +/- 3 months.
  As above.

SECONDARY OUTCOMES:
Tumour multiplicity | End of treatment at 24 months +/- 1 month
  The number of colorectal neoplasia (both benign and malignant tumors) per patient will be tested between groups by an analysis of variance, adjusting for country and history of cancer before randomization. In case of non-normally distributed residuals a suitable transformation to achieve normal distribution is considered. It will be tested whether 5-ASA (low- and high-dose together) reduces the number of any colorectal neoplasia (both benign and malignant tumors; tumor multiplicity) compared to placebo in LS patients at the end of treatment and end of study. Advanced adenomas are defined by a diameter above 1 cm villous or tubulo-villous histology or high grade dysplasia.
Tumour progress | End of treatment at 24 months +/- 1 month
  The tumor progress in 4 ordered stages will be tested between groups stratified for country and history of cancer before randomization.
  It will be tested whether 5-ASA reduces tumor progression (compared 4 ordinal stages: no colorectal neoplasia / non-advanced adenoma / advanced adenoma / carcinoma) compared to placebo in LS patients at the end of treatment and end of study. Advanced adenomas are defined by a diameter above 1 cm villous or tubulo-villous histology or high grade dysplasia.
Treatment effects | End of treatment at 24 months +/- 1 month
  The dependence of treatment effects on history of colorectal cancer, sex and patients age will be assessed by modelling interactions between these factors and treatment in the corresponding regression models.
  If differences between 5-ASA effects and placebo effects on the occurrence of colorectal neoplasia, tumor multiplicity or tumor progression depend on the history of colorectal cancer, sex and patients age will be investigated.
Significant findings & illnesses - adverse events | End of treatment at 24 months +/- 1 month
  Safety data are described and compared between groups in an exploratory manner to determine the safety concerning 5-ASA in LS patient. Therefore significant findings/illnesses, reported after the start of the study and which meet the definition of an AE, will be recorded in the CRF.
  Intention to treat set: This analysis set includes subjects who were randomized (and received at least one dose study drug). This analysis set will be chosen for safety assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Sofie Backman, MD PhD, Principal Investigator — Karolinska Institutet
Locations (8):
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Hvidovre Hospital, Hvidovre
- Sweden (6):
  - Sahlgrenska University Hsospital, Gothenburg, Gothenburg
  - Skåne University Hospital, Malmo, Skåne County
  - Ersta Hospital/Ersta Diakoni, Stockholm
  - Karolinska University Hospital, Stockholm
  - Norrland University Hospital, Umeå
  - Akademiska hospital, Uppsala

REFERENCES:
- [Derived] Backman AS, Frank A, Lindberg LJ, Ljungman D, Silander G, Gustafsson RJ, Bozso T, Schmidt PT, Ingre M, Mittlbock M, Lowbeer C, Marsal J, Lindblom A, Tham E, Therkildsen C, Gasche C; International MesaCAPP Study Group. Mesalamine for Colorectal Cancer Prevention Programme in Lynch syndrome (MesaCAPP): a multicentre, multinational, randomised, two-arm, double-blind, phase II clinical study with mesalamine or placebo in carriers with Lynch syndrome - a study protocol. BMJ Open. 2025 Nov 9;15(11):e100082. doi: 10.1136/bmjopen-2025-100082. PMID 41213710